CLINICAL TRIAL: NCT05796284
Title: Effects of Breast Tenderness Relief Intervention During the Late Pregnancy on the Parturients' Breast Engorgement, Lactation, Breastfeeding, Maternal Competence, and Stress
Brief Title: Effects of Breast Intervention During the Late Pregnancy on the Parturients' Breast Engorgement,Maternal Competence,and Stress
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Hsiang-Yun Lan, Associate Professor, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: C202205166
Record Dates: First submitted 2023-02-16; First posted 2023-04-03 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Breastfeeding; Pregnancy Related; Efficacy, Self
Keywords: breast tenderness relief intervention; breast engorgement; breastfeeding; maternal efficacy
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breast pressure relief intervention at the end of pregnancy (Experimental): The "Breast Compression Intervention at the End of Pregnancy" group is expected to start after the 36th week of pregnancy and continue until three months after delivery. In addition to routine care, breast relaxation methods of different intensities during pregnancy and postpartum will be provided in stages.
  Interventions: Behavioral: Breast pressure relief intervention at the end of pregnancy; Other: Routine care
- Routine care group (Active Comparator): Cases in the routine care group receive routine prenatal care and guidance during weekly outpatient checkups, and routine postpartum care and guidance after delivery, including breastfeeding posture and skills, hand expression, and breast milk storage methods, etc.
  Interventions: Other: Routine care

INTERVENTIONS:
Behavioral: Breast pressure relief intervention at the end of pregnancy — When teaching pregnant women, the researchers will use tablet computers and models to explain the operation of breast combing and acupressure one-on-one, and use the model to demonstrate. Emphasis on breast grooming during pregnancy, twice a day, once in the morning and evening, 5 minutes on one breast each time, 10 minutes on both sides; strengthen breast grooming and acupressure after delivery. The first breast combing, 5 minutes on one breast each time, and 10 minutes on both sides 4 to 6 times a day. After combing, according to expert advice, massage the 6 acupoints around the breast for 5-10 seconds, and then use hand expressing or breastfeeding to discharge the milk .
  Arms: Breast pressure relief intervention at the end of pregnancy
Other: Routine care — Cases in the routine care group received routine prenatal care and guidance during weekly outpatient checkups, and routine postpartum care and guidance after delivery.

SUMMARY:
The study purpose is to examine the effects of breast tenderness relief intervention during the late pregnancy on the parturients' breast engorgement, lactation, breastfeeding, maternal competence, and stress.

DETAILED DESCRIPTION:
Background:

Maternal and child health is an important global health issue. Breast milk is the best food for infants and has many benefits for both mothers and infants. However, the breastfeeding rate in Taiwan has not increased but decreased in recent years. Breast engorgement and hypogalactia often cause distress for many women, and lead to stress and abandonment of breastfeeding, which in turn affects the achievement of motherhood. Therefore, nurses should provide support interventions for parturients early.

Methods:

This study is a two-years, prospective randomized controlled trial, and will adopt a longitudinal repeated-measures design. Convenience sampling will be used to recruit 180 pregnancy and postpartum women in the obstetrics clinic and postpartum ward of a medical center. The participants will be randomly assigned into two conditions (routine care and the breast tenderness relief intervention condition). The intervention will be provided to the participants from the 36th week of pregnancy until three months after delivery. Questionnaires, and biological measurements will be used to collect data. The outcome variables include the degree of breast engorgement, lactation, breastfeeding, maternal competencies, and stress. In addition, those data will be collected at the 36th and 38th week of pregnancy, three days, six weeks, and twelve weeks after childbirth. It is expected to analyze the research results with generalized estimation equation method.

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy pregnant women over 20 years old, without mental illness, and the number of pregnancy weeks has reached 36 weeks; 2. Full term production; 3. Literate or able to communicate in Chinese and Taiwanese; 4. After explaining, agree to participate in the research, sign the consent form, and accept long-term follower

Exclusion Criteria:

1. Pregnant women with a history of smoking, alcohol, and drug abuse;
2. Pregnant women have mental illness;
3. Maternal complications during childbirth or postpartum, such as: postpartum hemorrhage, infection, etc.;
4. Newborns with congenital abnormalities and major diseases;
5. Pregnant women who are unable or unwilling to breastfeed due to illness or other factors;
6. Refuse to accept breast compression intervention will be excluded from participating in the study

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
breast engorgement | Change from Baseline breast engorgement at 12 weeks after delivery.
  the late pregnancy on the parturients' breast engorgement
The volume and speed of lactation | Change from Baseline lactation at 12 weeks after delivery.
  the late pregnancy on the parturients' lactation
Breastfeeding Self-efficacy Scale Short Form | Change from Baseline Breastfeeding Self-efficacy at 12 weeks after delivery.
  the late pregnancy on the parturients' breastfeeding
Parental Self-efficacy Scale | Change from Baseline Parental self-efficacy at 12 weeks after delivery.
  the late pregnancy on the parturients' maternal competence
Perceived Stress Scale | Change from Baseline Perceived Stress Scale at 12 weeks after delivery.
  late pregnancy on the parturients' stress

CONTACTS AND LOCATIONS:
Locations (1):
- National defense medical center, Taipei, Taiwan